CLINICAL TRIAL: NCT07276178
Title: Reliability of the Turkish Version of the Scoliosis Caregiver Response and Emotional Scale (SCaRES) Questionnaire
Brief Title: Reliability of the Scoliosis Caregiver Response and Emotional Scale (SCaRES) Questionnaire
Status: Not yet recruiting | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba GÖNEN, Assist. Prof. Dr., Hasan Kalyoncu University
Other Study IDs: 2025/126
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Scoliosis Idiopathic; Scoliosis Idiopathic Adolescent; Caregiver Anxiety
Keywords: Scoliosis Idiopathic Adolescent; Reliability; Caregiver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Scoliosis Caregiver Group: Demographic information of caregivers who met the study criteria will be recorded at the beginning of the study. In this study, written permission was obtained from the authors of the original scale to establish the reliability and psychometric properties of the Turkish version of the Scoliosis Caregiver Response and Emotional Survey. The scale was first translated into Turkish by two independent translators, and the translations were combined and synthesized by experts (physiotherapy/rehabilitation specialists and a linguist). The resulting Turkish version was back-translated into English by an independent translator and checked for consistency with the original text. The Scoliosis Caregiver Response and Emotional Scale (SCaRES) is a specific scale developed to measure the emotional and behavioral responses of parents or primary caregivers of children or adolescents with scoliosis to the treatment process. The scale assesses dimensions such as stress, anxiety, social limitations, and

SUMMARY:
The aim of this study is to examine the psychometric properties of the Turkish version of the Scoliosis Caregiver Response and Emotional Scale (SCaRES) questionnaire; to evaluate the reliability of the Turkish form and to ensure its usability in clinical and research fields.

DETAILED DESCRIPTION:
dependent on the involvement of families and caregivers. The emotional burden, stress, anxiety, and social limitations experienced by caregivers during the treatment process can indirectly affect both the individual's quality of life and the success of the patient's treatment. Therefore, objectively assessing the emotional and psychosocial impact experienced by caregivers of individuals with scoliosis is crucial for planning appropriate supportive interventions. The Scoliosis Caregiver Response and Emotional Scale (SCaRES), developed for this purpose, is a specific measurement tool that assesses emotional and behavioral responses to the treatment process in caregivers of individuals with scoliosis. Validity and reliability studies are required for the scale's use in different cultures and languages. Cultural differences, linguistic shifts, and healthcare system dynamics limit the scale's direct translation. Therefore, developing a Turkish version of the SCaRES is crucial for validly and reliably assessing the psychosocial burden experienced by caregivers in Turkish society. The aim of this study was to examine the psychometric properties of the Turkish version of the Scoliosis Caregiver Response and Emotional Scale (SCaRES) and to assess its reliability and ensure its usability in clinical and research settings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are an adult (parent or primary caregiver) responsible for the care of an individual diagnosed with scoliosis between the ages of 10 and 18.
* Individuals who are able to read and understand Turkish.
* Individuals who are actively involved in the child's treatment process (e.g., use of a brace, exercise program, follow-up appointments).
* Individuals who volunteer to participate in the study.

Exclusion Criteria:

* Participants whose children have a history of other comorbidities (neurological, etc.),
* Children whose children have a history of spinal surgery,
* Individuals who do not have an active role in the care process (e.g., parents who only provide financial support),
* Caregivers with intellectual disabilities, serious psychiatric diagnoses, or cognitive impairments that limit communication,
* Participants with incomplete or invalid survey forms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample population consists of individuals who volunteered for the study and met the inclusion criteria, who had no history of other comorbidities in their children, a positive neurological examination, or previous spinal surgery. Convenience sampling will be used in sample selection.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Scoliosis Caregiver Affect and Emotional Questionnaire Turkish Version | through of the study, average 6 months
  The Scoliosis Caregiver Response and Emotional Scale (SCaRES) is a specific scale developed to measure the emotional and behavioral responses of parents or primary caregivers of children or adolescents with scoliosis to the treatment process. The scale assesses aspects such as stress, anxiety, social limitations, and psychosocial burden experienced during the caregiving process. The SCaRES scale consists of 18 items. Each item is scored on a Likert-type scale of 1- Never, 2- Rarely, 3- Often, and 4- Always. The total scale score indicates the caregiver's level of impact on the treatment process. A higher score indicates a greater level of emotional and behavioral impact on the caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba GÖNEN, Asisst. Prof. Dr., Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Motyer G, Dooley B, Kiely P, Fitzgerald A. Parents' information needs, treatment concerns, and psychological well-being when their child is diagnosed with adolescent idiopathic scoliosis: A systematic review. Patient Educ Couns. 2021 Jun;104(6):1347-1355. doi: 10.1016/j.pec.2020.11.023. Epub 2020 Nov 25. PMID 33280964
- [Result] Campbell M, Matsumoto H, St Hilaire T, Roye BD, Roye DP, Vitale MG. Burden of care in families of patients with early onset scoliosis. J Pediatr Orthop B. 2020 Nov;29(6):567-571. doi: 10.1097/BPB.0000000000000711. PMID 31895294
- [Result] Shi Z, Mao Z, Xue S, Chen G, Li S. What is the relationship between health-related quality of life among scoliosis patients and their caregiver burden? A cross-sectional study in China. BMC Psychol. 2023 Oct 19;11(1):346. doi: 10.1186/s40359-023-01375-0. PMID 37858224
- [Result] Li C, Miao J, Gao X, Zheng L, Su X, Hui H, Hu J. Factors Associated with Caregiver Burden in Primary Caregivers of Patients with Adolescent Scoliosis: A Descriptive Cross-Sectional Study. Med Sci Monit. 2018 Sep 15;24:6472-6479. doi: 10.12659/MSM.909599. PMID 30218532
- [Result] Altaf F, Gibson A, Dannawi Z, Noordeen H. Adolescent idiopathic scoliosis. BMJ. 2013 Apr 30;346:f2508. doi: 10.1136/bmj.f2508. No abstract available. PMID 23633006
- [Result] Weinstein SL, Dolan LA, Cheng JC, Danielsson A, Morcuende JA. Adolescent idiopathic scoliosis. Lancet. 2008 May 3;371(9623):1527-37. doi: 10.1016/S0140-6736(08)60658-3. PMID 18456103
- [Result] Zaina F, Ferrario I, Bakhsh HR, Donzelli S, Negrini S. SCaRES - scoliosis caregiver response and emotional scale: a Rasch-validated questionnaire to measure the psychological impact of children's scoliosis on their parents. Eur Spine J. 2025 Nov;34(11):5224-5231. doi: 10.1007/s00586-025-08983-x. Epub 2025 Jun 21. PMID 40542837